CLINICAL TRIAL: NCT05564793
Title: ICONIC-M: Improving CRT Outcome With Non-Invasive Cardiac Mapping. A Multicenter Randomized Controlled Study To Assess Patient Response to CRT Comparing ECGI Map Guided Left Ventricular Lead Placement With Empirical Lead Placement
Brief Title: Improving CRT Outcome With Non-Invasive Cardiac Mapping
Acronym: ICONIC-M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EP Solutions SA (Industry)
Collaborators: QserveCRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DCR013-22
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Cardiac Resynchronization Therapy; Left Bundle Branch Block
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: A multicenter randomized controlled study to assess patient response to cardiac resynchronization therapy comparing ECGI map guided left ventricular lead placement with empirical lead placement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): The CRT device is implanted according to clinical practice, without pre-implantation planning. The outcome of the procedure is assessed via echography as per clinical practice.
  In addition to clinical practice, the subjects are required to fill in a quality-of-life questionnaire and are subject to an ECG mapping procedure with the Amycard 01C device, including non-contrast CT, to assess the distance between left ventricular lead placement and the latest electrical activation site in the absence of planning information.
  Interventions: Device: Post-implantation assessment
- Active (Experimental): A pre-implantation ECG mapping with the Amycard 01C device, including CT, is performed prior to the CRT device implantation. The resulting target area for the left ventricular lead placement is communicated to the implanting physician, who will attempt to reach a point close to the target, using the available venous access. At six-month follow-up, response to the therapy is assessed using echocardiography, and a second ECG mapping with Amycard 01C is performed, to assess the distance between actual implantation site and target in the presence of pre-implantation planning information.
  Interventions: Device: Pre-implantation planning; Device: Post-implantation assessment

INTERVENTIONS:
Device: Pre-implantation planning — ECGi mapping using the CE marked Amycard 01C device and a contrast enhanced CT
  Other Names: ECGI mapping
  Arms: Active
Device: Post-implantation assessment — ECGi mapping using the CE marked Amycard 01C device and a non-contrast CT
  Other Names: ECGI mapping

SUMMARY:
The ICONIC-M study is a multicenter randomized controlled study to assess patient response to CRT comparing ECGI map guided left ventricular lead placement with empirical lead placement.

The hypothesis of the investigation is to demonstrate that CRT LV lead implantation guided by a map obtained with the Amycard 01C System and showing LV Latest Electrical Activated Site (LEAS) in combination with a CT cardiac venogram improves CRT outcome. An improved CRT outcome is defined as a ≥30% increase in LVESVi reduction compared to empiric CRT LV lead implantation.

The sample size will be 136 in the Control arm and 194 in the Active arm. A total of 330 subjects.

The study follows an adaptive design, in where one interim analysis at 70% enrollment will be performed. The sponsor may stop enrollment when either one of the following conditions apply:

* Statistical significant difference between groups in the primary endpoint has been reached confirming a difference in reduction of the LVESVi of ≥30% in the Active arm compared to the Control arm
* There is no trend or reason to believe statistical significance will be reached with a higher sample size.

Statistical significance (primary endpoint) is reached at interim (70%) or at total (100%) of enrollment with a significance value P lower than 0.025.

DETAILED DESCRIPTION:
The study is conducted at European sites as a Post-Market Clinical Follow-Up study of a CE marked device (Amycard 01C). Its aim is to strengthen clinical evidence by assessing whether the use of this device for CRT planning improves clinical outcome in a statistically significant number of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Appropriately signed and dated informed consent.
2. Age ≥18 years at time of consent.
3. Received optimal medical therapy for HF for at least 3 months before screening
4. Patient in sinus rhythm at the time of screening fulfilling Class I or IIa criteria per ESC CRT guidelines 2013 .
5. Patient is intended for placement of a CRT device with biventricular (BiV) pacing.

Exclusion Criteria:

1. Previous cardiac pacemaker/CRT/ICD implantation
2. Acute diseases or exacerbations of chronic diseases (as per the investigator's discretion)
3. Contraindications to CT scanning
4. Contraindications to body surface ECG mapping: (ongoing wound healing on the chest (e.g. recent surgery), skin diseases, allergic reactions to surface mapping electrodes and medical band-aid)
5. Pregnant, or subjects planning to become pregnant within 6 months after signing informed consent (a documented negative pregnancy test (serum or blood) is required for women of childbearing potential)
6. Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority, are excluded from the study population

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of left ventricular end-systolic volume index (LVESVi) | 6 months post CRT implantation
  Reduction versus baseline of LVESVi as measured by transthoracic echocardiography

SECONDARY OUTCOMES:
Successfully placed LV leads | 6 months post CRT implantation
  Rate of successfully placed LV leads in the control and active arms
Correctly predicted distance between latest activation site and LV lead | 6 months post implantation
  Rate of correctly predicted distance between the latest electrical activation site, as identified with Amycard 01C, and the LV lead, as identified on CT

OTHER OUTCOMES:
Clinical Composite Score | 6 months post CRT implantation
  Clinical composite score consisting of Quality of life questionnaire, mortality rate and heart failure hospitalization rate
ECGi acquisition procedural failure rate | 6 months post CRT implantation
  Rate of unsuccessful ECGi mapping procedures using the Amycard 01C device
Subgroup analysis | 6 months post CRT implantation
  Subgroup analysis including stratification based on various conditions or habits (ischemia, diabetes, smoking, pulmonary disease, impaired right ventricular function, etc)
Shift of Latest Electrical Activation Site | 6 months post CRT implantation
  Degree of shift of the latest electrical activation site, as identified using the Amycard 01C device, between baseline and the six-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Varma, Prof., Principal Investigator — The Cleveland Clinic
Locations (11):
- Netherlands (5):
  - Amsterdam University Medical Center, Amsterdam
  - Groningen University Medical Center, Groningen
  - Leids Universitair Medical Center, Leiden
  - Maastricht University Hospital, Maastricht
  - Utrecht University Medical Center, Utrecht
- Hospital da Luz, Lisbon, Portugal
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm
- United Kingdom (3):
  - Bart's Hospital, London
  - King's College, London
  - Oxford University Hospital, Oxford